CLINICAL TRIAL: NCT05621499
Title: The Safety and Efficacy of HAIC or Lenvatinib Combined With Sintilimab as a Neoadjuvant Therapy for High Recurrence Risk Resectable Stage IB Solitary Hepatocellular Carcinoma: a Prospective, Randomized, Two Cohort, Exploratory Study
Brief Title: HAIC or Lenvatinib Combined With Sintilimab for High Recurrence Risk Resectable Solitary Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C20221044
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group1 (Experimental): HAIC
  Interventions: Drug: HAIC
- experimental group 2 (Experimental): Lenvatinib+Sintilimab
  Interventions: Drug: Sintilimab; Drug: Lenvatinib

INTERVENTIONS:
Drug: HAIC — Oxaliplatin 85 mg/m2, LV 400 mg/ m2, 5-FU 400 mg/m2 bolus and then 2400 mg/m2 as 46h continuous infusion，Q3W，a total of 2 cycles
  Arms: experimental group1
Drug: Sintilimab — 200mg，iv，d1，q3w，a total of 3 cycles
  Other Names: IBI308
  Arms: experimental group 2
Drug: Lenvatinib — 12 or 8mg/kg，po，qd，a total of 3 cycles
  Arms: experimental group 2

SUMMARY:
To evaluate the safety and efficacy of HAIC or Lenvatinib combined with Sintilimab as a neoadjuvant therapy for high recurrence risk resectable stage IB solitary hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to join the study and signed the informed consent form
* Aged 18-75, male or female
* ECOG PS score 0-1
* Child Pugh liver function Grade A
* Histopathology confirmed primary hepatocellular carcinoma (HCC) and the lesion met the indications for surgical resection in the Diagnostic and Therapeutic Norms for Primary Liver Cancer (2022)
* According to the investigator's assessment, there are the following high recurrence risk factors, Stage Ⅰ b: solitary tumor, with the largest diameter > 5cm
* At least one measurable lesion according to RECIST 1.1 (measurable lesion CT/MRI scan length diameter ≥ 10mm or lymph node lesion CT/MRI scan short diameter ≥ 15mm, and measurable lesion has not received radiotherapy, cryotherapy and other local treatments)
* Expected life ≥ 6 months
* Functions of important organs shall meet the following requirements (excluding the use of any blood component and cell growth factor within 14 days) Neutrophils ≥ 1500/mm3Platelet count ≥ 60,000/mm3Hemoglobin ≥ 5.6 mmol/L (9 g/dL); Serum creatinine (SCR) ≤ 1.5 times the upper limit of normal value (ULN) or creatinine clearance ≥ 50 ml/min (Cockcroft Gault formula); Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN); The level of AST or ALT ≤ 2.5 times the upper limit of normal value (ULN); Urine protein<2+; If urinary protein ≥ 2+, the 24-hour urine protein quantitative display must be ≤ 1g
* Normal coagulation function, no active bleeding and thrombosis disease

  1. International normalized ratio INR ≤ 1.5 × ULN；
  2. Partial thromboplastin time APTT ≤ 1.5 × ULN；
  3. Prothrombin time PT ≤ 1.5ULN;
* Women of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the medication period and within 6 months after the end of medication; If the serum or urine pregnancy test was negative within 7 days before the study included, and the patient must be a non lactating patient, the male should agree to use contraception during the study period and within 6 months after the end of the study period
* The subjects had good compliance and cooperated with follow-up.

Exclusion Criteria:

* Previously received radiotherapy, chemotherapy, concurrent radiotherapy and chemotherapy or other targeted therapies
* Known hepatobiliary cell carcinoma, sarcomatoid HCC, mixed cell carcinoma and fibrolamellar cell carcinoma; Have other active malignant tumors except HCC within 5 years or at the same time
* Patients with hypertension who cannot be well controlled after antihypertensive drug treatment (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg); Previous hypertension crisis or hypertensive encephalopathy
* Patients had other malignant tumors in the past or at the same time (except cured skin basal cell carcinoma and cervical carcinoma in situ);
* Patients who had been treated with Sintilimab or other PD-1/PD-L1 inhibitors in the past could not be included; Known hypersensitivity to macromolecular protein preparations or any excipients of Sintilimab or lenvatinib
* Patients have any active autoimmune diseases or have a history of autoimmune diseases (Including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; Patients with vitiligo or asthma in childhood has completely alleviated, without any intervention after adulthood can be included; Patients with asthma requiring medical intervention of bronchodilators cannot be included)
* Patients who are using immunosuppressive agents, or systemic or absorbable local hormone to achieve immunosuppressive purpose (Dose>10mg/day prednisone or other equivalent therapeutic hormones) and continue to use them within 2 weeks before enrollment
* Ascites or pleural effusion with clinical symptoms and requiring therapeutic puncture or drainage
* There are clinical symptoms or diseases of the heart that are not well controlled, such as:

  1. Heart failure above NYHA level 2
  2. Unstable angina pectoris
  3. Myocardial infarction occurred within 1 year
  4. Clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention
* Patients having gastrointestinal diseases such as esophageal varices, active gastric and duodenal ulcers, ulcerative colitis, portal hypertension, or active bleeding from tumors that have not been removed, or other conditions that may cause gastrointestinal bleeding and perforation as determined by the investigator at present (within 3 months)
* Serious bleeding (>30 ml bleeding within 3 months), hemoptysis (>5 ml fresh blood within 4 weeks) or thromboembolism (including stroke and/or transient ischemic attack) occurred in the past or present
* Patients with active infection or fever of unknown origin>38.5℃during the screening period and before the first administration (according to the judgment of the investigator, subjects with fever due to tumor can be included)
* Patients with past or current objective evidence of pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, and severe impairment of pulmonary function
* Patients with congenital or acquired immune deficiency, such as HIV infection, or active hepatitis (transaminase does not meet the inclusion criteria: HBV DNA ≥ 10e4/ml; HCV RNA ≥ 10e3/ml); Chronic hepatitis B virus carriers with HBV DNA<2000 IU/ml (<10e4 copies/ml) receive antiviral treatment at the same time during the trial can be included
* Live vaccine may be inoculated less than 4 weeks before the study medication or during the study period
* Known history of abuse of psychotropic substances, alcohol abuse or drug abuse
* Conditions should be excluded according to the judgment of the investigator, for example, according to the judgment of the investigator, the patient has other factors that may lead to the forced termination of the study, such as other serious diseases requiring combined treatment, serious laboratory examination abnormalities, and family or social factors, which may affect the safety of the subject, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
1-year DFS rate | up to 1 years
  To evaluate the 1-year disease free survival rate of neoadjuvant treatment with HAIC or Lenvatinib combined with Sintilimab for of high recurrence risk resectable stage IB solitary hepatocellular carcinoma

SECONDARY OUTCOMES:
Incidence of microvascular invasion | Up to 3 years
  Defined as proportion of patients with microvascular invasion
Pathological complete response rate (pCR) | up to 1 years
  Defined as proportion of patients who have a best response of pCR
Objective response rate | Up to 1 years
  Defined as proportion of patients who have a best response of CR or PR
2-year DFS rate | Up to 3 years
  To evaluate the 2-year disease free survival rate of neoadjuvant treatment with HAIC or Lenvatinib combined with Sintilimab for of high recurrence risk resectable stage IB solitary hepatocellular carcinoma
2-year OS rate | Up to 3 years
  To evaluate the 2-year overall survival rate of neoadjuvant treatment with HAIC or Lenvatinib combined with Sintilimab for of high recurrence risk resectable stage IB solitary hepatocellular carcinoma
Adverse Events (AEs) | Up to 3 years
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0 and complications of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China